CLINICAL TRIAL: NCT06244524
Title: Exploring the Influence of Elevated Indoor CO2 Levels on Allergic Skin Disorders
Brief Title: Exploring the Influence of Elevated CO2 on Allergic Skin
Acronym: EICO2AS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Swiss Institute of Allergy and Asthma Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EICO2AS
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Affects of Elevated Indoor CO2

STUDY DESIGN:
Intervention Model Description: The recruited healthy donors will be randomly distributed into ventilated or closed bedrooms. We will assess the epithelial barrier function on their forearm by electrical impedance spectroscopy before and after 8 hours of sleep in each bedroom. The level of CO2 in the bedrooms will be monitored. In addition, the skin biopsy samples will be collected from fore arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Well-ventilated bedroom (No Intervention): The participants will stay and sleep for eight hours in a well-ventilated bedroom.
- Non-ventilated bedroom (Experimental): The participants will stay and sleep for eight hours in a closed bedroom.
  Interventions: Other: High indoor CO2 exposure

INTERVENTIONS:
Other: High indoor CO2 exposure — The participants will stay and sleep for eight hours in a closed bedroom.
  Arms: Non-ventilated bedroom

SUMMARY:
The goal of this clinical trial is to investigate the impact of elevated indoor CO2 levels on skin barrier function and inflammation in healthy adults. The main questions it aims to answer are:

How do increased indoor CO2 levels contribute to type 2 inflammation and barrier dysfunction in human skin? What is the demonstrable impact of high CO2 exposure on the human skin barrier and transcriptome? Participants will be exposed to controlled levels of CO2 in either well-ventilated or non-ventilated (closed) bedrooms.

We will evaluate epithelial barrier function by electrical impedance spectroscopy (EIS), collect skin biopsy samples, and investigate the change induced by high indoor CO2 exposure. Healthy adults meeting the inclusion criteria will be included and those with chronic skin conditions, allergies, or recent systemic therapy will be excluded.

Researchers will compare participants exposed to elevated CO2 levels in closed bedrooms with those in well-ventilated bedrooms to determine if skin barrier integrity and transcriptome variations are observed.

DETAILED DESCRIPTION:
1. Core Message:

   Elevated indoor CO2 levels in closed rooms may contribute to skin barrier dysfunction and inflammation. Understanding the impact of increasing CO2 on the skin is essential to public health.
2. Supporting Information:

   Atopic dermatitis (AD) affects a significant population, and indoor CO2 levels are rising in the bedroom.

   Preliminary studies demonstrate the association between CO2 exposure and skin barrier dysfunction.

   Skin barrier functions can be assessed by electrical impedance spectroscopy (EIS) in vivo.
3. Key Points:

   Scientific Question: Investigate how increased indoor CO2 levels contribute to type 2 inflammation and barrier dysfunction in human skin.

   Proposed Intervention: Controlled human skin CO2 exposure experiments in well-ventilated vs. non-ventilated (closed) bedrooms.

   Scientific Basis: Preliminary studies have shown that elevated CO2 levels in closed spaces and validate EIS as a reliable assessment tool for skin barrier integrity assessment.
4. Objectives:

   Hypothesis: Elevated indoor CO2 affects skin homeostasis and barrier function. Primary Objective: Demonstrate the impact of high CO2 exposure on the human skin barrier and transcriptome.
5. Study Population and Procedures:

   Inclusion criteria: Healthy adults aged 18-65. Exclusion criteria: Individuals with chronic skin conditions, allergies, or recent systemic therapy.

   Recruitment through ongoing processes and physician referrals. Informed consent emphasizes voluntary participation and the right to withdraw.
6. Statistics and Methodology:

   Sample size: 50 participants to detect meaningful differences. Intervention: Participants will be randomly assigned to well-ventilated or non-ventilated (closed) bedrooms groups. The researcher will evaluate epithelial barrier by electrical impedance spectroscopy at 0h (before the exposure) and 8h (after the exposure).

   After exposure, the skin biopsy will be collected from the epithelial barrier measurement site.

   Statistical methods: Mann-Whitney U test and t-test for data analysis.
7. Regulatory Aspects and Safety:

   Compliance with Declaration of Helsinki, ICH-GCP, and local regulations. Immediate reporting of Adverse Events (AEs). Annual safety reports and notification of safety measures.
8. Quality Control and Data Protection:

   Measures include personnel training, SOPs, double data entry, and regular reviews.

   Data is handled with discretion, identified by unique participant numbers, and stored securely for 10 years.
9. Monitoring and Registration:

   SIAF and UZH will conduct monitoring; participants visit these sites for assessments.

   This study will be registered with the Swiss National Clinical Trial Portal (SNCTP via BASEC) and ClinicalTrials.gov.
10. Funding / Publication / Declaration of Interest:

Funding from Pathway Global Grant (Sanofi) and SciBase. Commitment to transparency, open science, and conflict-free reporting. Multicentre collaboration between SIAF and Swiss Dermatology Clinic.

ELIGIBILITY:
Inclusion Criteria:

The study population will consist of healthy adult volunteers; 1. age between18 and 65 years, 2. Generally healthy and able to provide written informed consent.

The choice of healthy adult volunteers without pre-existing skin conditions on site or allergies against tested products is justified.

Exclusion Criteria:

1. Severe dermatitis, eczema, psoriasis, or other chronic skin conditions.
2. History of hypersensitivity or allergies to tested product ingredients.
3. Current or recent systemic therapy for a skin condition in the past six months.
4. Pregnant or breastfeeding individuals.
5. Use of investigational drugs or participation in another trial in the last 30 days.
6. History of skin cancer or malignancies in the study area.
7. Significant sunburn, open wounds, or active skin infections in the study area.
8. Any medical condition that, per the investigator, might compromise safety or confound results.
9. Inability to follow study instructions or attend required clinic visits.
10. Gender Balance: To ensure gender balance, efforts will be made to recruit an equal number of male and female participants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Skin barrier evaluation | before (0 hour) and after 8 hours of sleep in ventilated or closed bedroom.
  We will measure skin barrier integrity by electrical impedance spectroscopy
Skin biopsy collection | After the electrical impedance measurment at 8 hours
  We will collect skin biopsy from the forearm that we measure electrical impedance

CONTACTS AND LOCATIONS:
Overall Officials: Yasutaka Mitamura, MD PhD, Principal Investigator — Swiss Institute of Allergy and Asthma Research

IPD SHARING:
Plan to Share IPD: No